CLINICAL TRIAL: NCT02608606
Title: Determining Equivalence Dose for Oral Versus Sublingual Administration of Tacrolimus in Hepatic Receptors
Acronym: FKosl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FKoral-sl
Record Dates: First submitted 2015-11-03; First posted 2015-11-20 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Evidence of Liver Transplantation; Effects of Immunosuppressant Therapy
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral administration of tacrolimus (No Intervention): Oral administration of tacrolimus (FK506) in the usal dose and measuring plasmatic levels at hours 0, 0.5, 1, 2, 3, 4 and 6. Measuring AUC.
- sublingual administration of tacrolimus (Active Comparator): sublingual administration of tacrolimus (FK506) in the dose that allows similar plasmatic level at time 0 compared with the oral administration, and measuring plasmatic levels at hours 0, 0.5, 1 , 2, 3 , 4 and 6. Measuring AUC.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — compared oral administration versus sublingual administration of tacrolimus.
  Other Names: FK506
  Arms: sublingual administration of tacrolimus

SUMMARY:
After liver transplantation one of the most important cost, for both patients and their health insurance system, is immunosuppressive drug therapy. Tacrolimus (FK 506) is considered the cornerstone of immunosuppressive therapy in solid organ transplantation. Oral administration is the usual route, however, sublingual (SL) administration has been recently reported. This method of administration avoids first pass metabolism and allows an alternative route after transplant surgery, particularly in those patients who should extend the period of fasting (prolonged intubation, ileus, etc). Interestingly, in some studies, the dose of tacrolimus SL required to maintain similar plasma concentrations compared with oral administration, is significantly lower, even up to 50%, which can result in considerable savings in short and long term. Among these studies, only one was conducted in liver recipients. This study suggest that SL administration of tacrolimus could allow to obtain similar concentrations compared with oral administration. The design of this study did not assess the existence of differences in the dose required and only included six patients.

DETAILED DESCRIPTION:
The patient will be scheduled fasting to liver transplant unit where the pharmacokinetic study was performed. After installation of the venous needle, blood samples will be collected on 4 ml tubes with EDTA as an anticoagulant at the following intervals of time in hours: 0 (immediately before the oral administration of tacrolimus); 0.5; 1.0; 1.5; 2; 4; 6; 9 and 12 h. post-dose. Once the blood samples taken, the tubes will be plugged, invest gently to mix with anticoagulant and stored at -20 ° C until analysis.

Subsequently, tacrolimus administration was change to sublingual route and dose was adjusted to obtain similar trough levels to those determined on per oral administration. The capsule be opened and its contents shall be deposited in the sublingual mucosa. To be ensure that drug will be absorted the patient will be instructed to insistently that after sublingual placement of the drug, should not swallow the capsule content for at least 15 minutes. The same pharmacokinetic study described for the oral route will be performed.

Breakfast will be administered 2 hours after ingesting the drug and lunch and dinner 6 and 10 hours after respectively. Fluid intake is discretionary.

ELIGIBILITY:
Inclusion Criteria:

* Outline of immunosuppression that includes tacrolimus dosing every 12 hours.
* Stable plasma levels of tacrolimus in 3 consecutive measurements.
* Stable blood tests: biochemical profile, creatinine and liver profile.
* Absence of treatment with drugs that have interaction with tacrolimus (antifungal and diltiazem) and use of grapefruit juice.
* Absence of active bacterial or viral infection and rejection episodes within 8 weeks prior.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Compare tacrolimus exposure using per oral and sublingual administration employing AUC (Area Under the Curve). | 30 days
  compared oral administration versus sublingual administration of tacrolimus

SECONDARY OUTCOMES:
Compare tacrolimus dose necessary to obtain similar trough levels employing per oral and sublingual administration | 30 days
  compared oral administration versus sublingual administration of tacrolimus

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Benitez, Hepatologist, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
The preliminary data from this trial will be presented at the AASLD Liver meeting in San Francisco in November 2015

REFERENCES:
- [Result] Agopian VG, Petrowsky H, Kaldas FM, Zarrinpar A, Farmer DG, Yersiz H, Holt C, Harlander-Locke M, Hong JC, Rana AR, Venick R, McDiarmid SV, Goldstein LI, Durazo F, Saab S, Han S, Xia V, Hiatt JR, Busuttil RW. The evolution of liver transplantation during 3 decades: analysis of 5347 consecutive liver transplants at a single center. Ann Surg. 2013 Sep;258(3):409-21. doi: 10.1097/SLA.0b013e3182a15db4. PMID 24022434
- [Result] Rabkin JM, Corless CL, Rosen HR, Olyaei AJ. Pharmacoeconomic study of tacrolimus-based versus cyclosporine-based immunosuppressive therapy following liver transplantation. Transplant Proc. 2001 Feb-Mar;33(1-2):1532-4. doi: 10.1016/s0041-1345(00)02585-9. No abstract available. PMID 11267411
- [Result] Collin C, Boussaud V, Lefeuvre S, Amrein C, Glouzman AS, Havard L, Billaud EM, Guillemain R. Sublingual tacrolimus as an alternative to intravenous route in patients with thoracic transplant: a retrospective study. Transplant Proc. 2010 Dec;42(10):4331-7. doi: 10.1016/j.transproceed.2010.09.126. PMID 21168693
- [Result] Reams BD, Palmer SM. Sublingual tacrolimus for immunosuppression in lung transplantation: a potentially important therapeutic option in cystic fibrosis. Am J Respir Med. 2002;1(2):91-8. doi: 10.1007/BF03256598. PMID 14720063
- [Result] Reams D, Rea J, Davis D, Palmer S. Utility of sublingual tacrolimus in cystic fibrosis patients after lung transplantation. J Heart Lung Transplant. 2001 Feb;20(2):207-208. doi: 10.1016/s1053-2498(00)00447-2. No abstract available. PMID 11250374
- [Result] Romero I, Jimenez C, Gil F, Escuin F, Ramirez E, Fudio S, Borobia A, Carcas A. Sublingual administration of tacrolimus in a renal transplant patient. J Clin Pharm Ther. 2008 Feb;33(1):87-9. doi: 10.1111/j.1365-2710.2008.00884.x. PMID 18211623
- [Result] Srinarong P, Pham BT, Holen M, van der Plas A, Schellekens RC, Hinrichs WL, Frijlink HW. Preparation and physicochemical evaluation of a new tacrolimus tablet formulation for sublingual administration. Drug Dev Ind Pharm. 2012 Apr;38(4):490-500. doi: 10.3109/03639045.2011.613075. Epub 2011 Sep 30. PMID 21961909
- [Result] Tsapepas D, Saal S, Benkert S, Levine D, Delfin M, Cremers S, Amann S, Dadhania D, Kapur S, Aull M. Sublingual tacrolimus: a pharmacokinetic evaluation pilot study. Pharmacotherapy. 2013 Jan;33(1):31-7. doi: 10.1002/phar.1149. PMID 23307542
- [Result] van de Plas A, Dackus J, Christiaans MH, Stolk LM, van Hooff JP, Neef C. A pilot study on sublingual administration of tacrolimus. Transpl Int. 2009 Mar;22(3):358-9. doi: 10.1111/j.1432-2277.2008.00779.x. Epub 2008 Oct 30. No abstract available. PMID 18980626
- [Result] Watkins KD, Boettger RF, Hanger KM, Leard LE, Golden JA, Hoopes CW, Singer JP. Use of sublingual tacrolimus in lung transplant recipients. J Heart Lung Transplant. 2012 Feb;31(2):127-32. doi: 10.1016/j.healun.2011.10.015. Epub 2011 Dec 16. PMID 22177691
- [Result] Nasiri-Toosi Z, Dashti-Khavidaki S, Nasiri-Toosi M, Khalili H, Jafarian A, Irajian H, Abdollahi A, Sadrai S. Clinical pharmacokinetics of oral versus sublingual administration of tacrolimus in adult liver transplant recipients. Exp Clin Transplant. 2012 Dec;10(6):586-91. doi: 10.6002/ect.2012.0032. Epub 2012 Jul 5. PMID 22770208